CLINICAL TRIAL: NCT00471510
Title: A Phase 2 Multicenter, Randomized, Placebo-Controlled, Parallel Group Dose-Ranging Study to Evaluate the Safety and Efficacy of Topical NEOSH101 in the Treatment of Androgenetic Alopecia in Men
Brief Title: Dose-Ranging Efficacy Study of Topical NEOSH101 to Treat Male Pattern Hair Loss
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neosil, Inc. (Industry)
Responsible Party: Andria Langeberg, MD, Vice President, Clinical Development, Neosil, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOSH101-CLIN-AGA004
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Androgenetic Alopecia
Keywords: androgenetic alopecia; male pattern hair loss; male pattern baldness; androgenetic alopecia or male pattern hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): NEOSH101 2%
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)
- 2 (Experimental): NEOSH101 1%
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)
- 3 (Experimental): NEOSH101 0.5%
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)
- 4 (Placebo Comparator)
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)

INTERVENTIONS:
Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101) — Study preparation (experimental, placebo comparator) will be applied to the scalp once daily for 16 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of three doses of topical NEOSH101 applied once-daily (qd) for 16 weeks in men with thinning hair in the top and center of the scalp (Norwood/Hamilton grades III-IV androgenetic alopecia). Four equally sized treatment groups (35 men each) will receive either NEOSH101 0.5%, NEOSH101 1.0%, NEOSH101 2.0% or placebo. A 12-week observation period will follow the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged 18 to 49 years, in general good health
* Norwood/Hamilton grades III - IV androgenetic alopecia, with thinning hair in the vertex area

Exclusion Criteria:

* Concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug
* Treatment with a systemic or locally acting medication which may interfere with the study objectives, such as minoxidil treatment in the 6 months prior to study day 1, finasteride treatment in the 12 months prior to study day 1, or treatment with other investigational hair growth products in the 6 months prior to study day 1

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Hair density, hair growth rate, hair diameter as measured using the Trichoscan method | 16 weeks application treatment period followed by 12 weeks observation period

SECONDARY OUTCOMES:
Assessment score of dermal tolerability | 16 weeks application treatment period followed by 12 weeks observation period
Physician's global assessment score | 16 weeks application treatment period followed by 12 weeks observation period

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gassmueller, MD, Principal Investigator — bioskin Institute for Dermatological Research and Development GmbH
Locations (1):
- bioskin Institute for Dermatological Research and Development GmbH, Hamburg, Germany